CLINICAL TRIAL: NCT01764074
Title: Brief Sleep Intervention for Suicide in Bipolar Disorder
Brief Title: Brief Sleep Intervention for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Instructor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRG-0-071-11
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Bipolar Disorder; Sleep Problems; Suicidal Thoughts
Keywords: Bipolar Disorder; Sleep Intervention; Suicide; Cognitive Behavioral Therapy; Sleep Quality
MeSH Terms: conditions — Bipolar Disorder; Parasomnias; Suicidal Ideation; Suicide; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brief Sleep Intervention (Experimental): Every participant in the study will complete a 3-session sleep intervention with a clinician to improve sleep problems such as insomnia or hypersomnia.
  Interventions: Behavioral: Brief Sleep Intervention

INTERVENTIONS:
Behavioral: Brief Sleep Intervention — Participants will meet with a therapist for three sessions to try to improve sleep problems (hypersomnia or insomnia, depending on the problems the participant has).

SUMMARY:
Individuals with bipolar disorder (BD) experience extreme mood swings, or episodes of depression and (hypo)mania. These episodes are associated with poor functioning, worse course of illness, and high rates of suicidality. It is estimated that between 25 to 65% of individuals with BD attempt suicide and 4 to 19% of individuals with BD eventually die by suicide. Sleep disturbance has been identified as a primary prodromal as well as causal symptom of mood episodes and recently, has been found to be associated with higher rates of suicidal ideation and behavior. Given the role that sleep may have in mood stability and suicidality in BD, it seems imperative to further understand the association of sleep and suicide and how sleep interventions may be useful to reduce suicidality in BD. Thus, the primary aim of this study is to use an innovative home sleep monitoring device, or the Embla, to examine the association of sleep and suicidality in adult outpatients with BD. The Embla is unique in that it is a non-invasive device that can characterize sleep profiles by measuring the degree of sleep fragmentation and percentage of rapid eye movement (REM) sleep. The study duration is five to six weeks such that patients wear the Embla device for Week 1, participate in a brief sleep intervention for suicide during Weeks 2 and 3, and 4, and then wear the Embla device for one more week (Week 5). This intervention consists of three, 60-min sessions and utilizes cognitive-behavioral therapy strategies (e.g., psychoeducation, cognitive re-structuring, problem solving, behavioral activation) to improve sleep disturbance. The investigators expect that individuals at study entry with more sleep disturbance (as measured by the Embla) will report more suicidal ideation and behaviors. The investigators also hypothesize that from pre- to post-intervention, individuals will report less sleep disturbance as well as suicidal ideation and behaviors. Data from this research has immediate and practical implications for providers and their patients as it the first examination of sleep phenotypes and suicide in a high risk population as well as to explore the association of improvements in sleep with suicidality.

DETAILED DESCRIPTION:
Bipolar disorder is characterized by episodes of depression as well as episodes of mania (abnormally high mood). Individuals with bipolar disorder experience high rates of suicidal ideation and behavior, with risk of death due to suicide estimated to be 20 times greater than the general population. Moreover, some research suggests that among individuals treated for bipolar disorder, approximately 40% will report a past suicide attempt. Other studies suggest that between 25 and 65% of patients with bipolar disorder will attempt suicide and that between 4 and 19% of these individuals will be successful. Among the DSM-IV-TR Axis I disorders, suicide appears to be the highest in bipolar disorder. Individuals with bipolar disorder have a greater likelihood of both current and past suicidal ideation if they have an anxiety disorder, have an earlier age of onset, or a more severe course of illness. Nevertheless, there is a continued need for information on the epidemiology and risk factors for suicidal ideation and behavior in this population.

Several studies have shown that sleep difficulties (i.e., insomnia, hypersomnia, poor sleep quality, and nightmares) are significantly associated with suicidal ideation, even after controlling for depression. These disturbances are well documented during episodes of depression and mania, but sleep disturbances have also been shown to persist during periods of relative mood stability. A common symptom in bipolar patients experiencing manic episodes is a reduced need for sleep, and several studies using polysomnography have identified decreased REM sleep latency in manic episodes. Utilizing self-report measures, studies of bipolar patients in depressive episodes have identified variable rates of hypersomnia and insomnia as common factors. However, research conducted using laboratory-based polysomnography during depressive episodes have reported disparate findings.

This proposal involves a test of a novel measure of sleep architecture in patients with bipolar disorder, using a newly available home sleep monitoring device called Embla (www.embla.com). This device sticks to the skin on the chest with standard EKG-adhesive stickers and captures electrocardiogram (EKG) during sleep. The Embla device also measures movement, snoring, body position, and light levels. The on-board storage allows 2-3 weeks of nightly recording. By using an unobtrusive and potentially informative measure of sleep architecture, this protocol will allow longitudinal, objective information about sleep disturbance to be compared with corresponding mood states in patients with bipolar disorder.

Overall, this protocol is investigating the relationship between suicidality and sleep disturbance as well as assessing whether a brief CBT intervention for sleep disturbance is associated with reduced suicidal ideation and/or behavior. Since research suggests that CBT is an effective adjunct treatment for reducing suicidality in this population, and that treatment for insomnia can improve sleep in individuals with bipolar disorder, the present research has important implications for the prevention and intervention of suicide in this vulnerable population. To the investigators knowledge, no investigations have looked at the effectiveness of CBT on both sleep and suicidality in bipolar disorder. Furthermore, while past research has relied almost exclusively on subjective reports of sleep, this study captures both subjective and objective measures of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Have a primary diagnosis of bipolar I or bipolar II disorder
* Have a reported sleep disturbance
* Have reported suicide ideation (thoughts)

Exclusion Criteria:

* Any known or active sleep disorder (such as sleep apnea)
* Any history of significant cardiac, pulmonary, neurological, hepatic, or renal disease
* Any history of malignancy, chemotherapy, or radiation
* Any skin condition that would prevent wearing the device
* Pregnancy
* Current or suspected sleep apnea
* Current use of certain medications including beta blockers
* Known diagnosis of atrial fibrillation
* Acute major depressive or manic episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
High Frequency Coupling (HFC) | 6 weeks
  High Frequency Coupling (HFC) is a measure of the portion of unstable versus stable sleep, and this is measured by the Embla device.
  HFC has been validated in a variety of circumstances, and correlates with cardiovascular and mental health outcomes(Thomas, 2006).
Modified Scale of Suicidal Ideation (MSSI) | 5 weeks
  The MSSI is a 19-item clinical research instrument designed to quantify and assess suicidal intention.
The Columbia-Suicide Severity Rating Scale (CSSRS) | 5 weeks
  The CSSRS records suicidal behavior on the basis of attempts, non-suicidal self-injurious behavior, interrupted attempts, aborted attempts, and preparatory acts or behaviors.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 5 weeks
  The MADRS is a 10-item clinician-rated scale to measure the overall severity of depressive symptoms.

OTHER OUTCOMES:
Percentage of rapid eye movement (REM) sleep | 5 weeks
Pittsburgh Sleep Quality Index (PSQI) | 5 weeks
  9-item self-rated questionnaire that measures sleep quality and sleep disturbance over the past month
Young Mania Rating Scale (YMRS) | 5 weeks
  The YMRS aims to quantify the degree of mania in patients who already have a diagnosis of BD and is the most widely studied instrument for mania

CONTACTS AND LOCATIONS:
Overall Officials: Louisa G Sylvia, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States